CLINICAL TRIAL: NCT00283946
Title: FK199B (Zolpidem MR Tablet) Phase III Clinical Study -A Double-blind, Group-comparison Study Using Zolpidem (Myslee) as a Comparative Drug in Patients With Insomnia -
Brief Title: A Double-blind, Group-comparison Study Using Zolpidem (Myslee) as a Comparative Drug in Patients With Insomnia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6199-CL-0007
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Initiation and Maintenance Disorders; Sleep Disorders
Keywords: zolpidem; sleep initiation and maintenance disorders Hypnotics and sedatives; double-blind study; comparative study
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Zolpidem MR
- 2 (Active Comparator)
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem MR — Oral
  Arms: 1
Drug: Zolpidem — Oral
  Other Names: Myslee
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of FK199B (Zolpidem MR Tablet) in patients with insomnia by a randomized, double-blind, group-comparison study using zolpidem (Myslee) as a comparative drug

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of nonorganic insomnia.
* Must be able to swallow tablets

Exclusion Criteria:

* Allergic reactions to zolpidem (Myslee)
* Serious cardiac disorders; Serious hepatic impairment; Serious renal diseases, etc.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 876 (Actual)
Dates: Start 2006-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Mean wake time after sleep onset during the double-blind period | 2 Weeks

SECONDARY OUTCOMES:
Mean total sleep time during the double-blind period | 2 Weeks
Mean number of nightly awakenings during the double-blind period | 2 Weeks
Mean sleep latency during the double-blind period | 2 Weeks
Patient impression during the double-blind period | 2 Weeks
Safety | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kansai Region
  - Kanto Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region